CLINICAL TRIAL: NCT06369857
Title: Pectopexy for Treatment of Apical Pelvic Organ Prolapse
Brief Title: Pectopexy for Apical Prolapse Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Lecturer of Obs& Gyn. Specialist of Urogynecology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPY
Record Dates: First submitted 2024-03-24; First posted 2024-04-17 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Case series study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pectopexy (Experimental): All operations will be performed with patient in loyd davies position, sterilization of the perineum then sterilization of the vagina.
  Evacuation of the bladder and examination under anesthesia is done.
  Skin incision through pfannenstiel one then incision of subcutaneous tissue, rectus sheath, separation of recti muscle and opening of parietal peritoneum.
  A polypropylene mesh (30×30 cm, Ethicon, Inc., Somerville, NJ) is cut to obtain two long arms (15-20 cm long) and a rectangular piece (4-7 cm wide). The mesh is fashioned and fixed over the dissected uterine isthmus and anterior part of the cervix with separated number 1 Prolene and number 1 Vicryl sutures.
  Peritoneal incision was made from the right round ligament toward the pelvic side wall .
  The mesh arm is grasped and laterally pulled out So the rectangular part of the mesh will be on the anterior part of the cervix The mesh arms are suspended and sutured to Pectineal liga peritoneum is closed over the mesh
  Interventions: Procedure: Pectopexy

INTERVENTIONS:
Procedure: Pectopexy — Suspension of apical organs

SUMMARY:
This study was designed to evaluate the efficacy of pectopexy for treatment of apical pelvic organ prolapse at follow up at 12 months. Investigator also evaluates complications, improvement of symptoms, quality-of-life outcomes and patient satisfaction with surgery.

Assessment of restoration of normal pelvic anatomy and lower urinary tract symptoms using transperineal ultrasound

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) substantially affects the quality of life (QOL) of women, with a global prevalence of 20% to 65% .Surgery is the major treatment option for patients with POP at POP Quantification (POP-Q) stage ≥II, especially after failure of conservative treatments . Apical pelvic organ prolapse is a common issue in Egypt with significant incidence rate due to many predisposing factors including increasing age, higher gravidity and parity (especially the number of vaginal births .

Apical support is the most important factor for the successful outcome of pelvic reconstruction surgery. Apical suspension can be performed transabdominally or transvaginally using native tissue or a synthetic mesh . Abdominal sacropexy is considered now the gold standard operation for treatment of apical pelvic organ prolapse . However , many intraoperative complication can occur including hemorrhage or transfusion or both occurred in 4.4% , intestinal injury or rectal injury in 1.6% (0.4% to 2.5%),and ureteral injury in 1.0% of cases. Postoperative complications include paralytic ileus in 3.6%.transient femoral nerve injury and vertebral osteomyelitis . Sacropexy also has a long steep learning curve .

Pectopexy has been in 2011 where synthetic mesh is fixed to the pectineal ligaments bilaterally.This surgery is presumed to have fewer complications because the surgical field is limited to the anterior pelvis, with a decreased risk of injury to the adjacent organs. The technique is suitable for surgeons seeking an attractive alternative for patients in a context of high morbidity and/or with difficult access to the promontory . However, adequate evidence to support this surgical option still needs further studies.

ELIGIBILITY:
Inclusion Criteria:

* Apical prolapse Stage 2-4 acc. to POP-Q system
* Uterine preservation or after hysterectomy
* Age > 18 years old.
* Sexually active or not.

Exclusion Criteria:

* Pregnancy or up to 6 months postpartum.
* Current Urinary tract infection proved by urine analysis or urine culture.
* Patient unfit for surgery.
* Previous suspension operations.
* Uncontrolled diabetic patients

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification stage | 6 , 12 months
  Stage 0 to stage 4

SECONDARY OUTCOMES:
Urinary Symptoms questionnaire | 6 , 12 months months
  Questions about urinary system before and after surgery
Bladder neck measurements using Transperineal US | 6 , 12 months
  Bladder neck height in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital, Asyut, Egypt